CLINICAL TRIAL: NCT05608681
Title: A Phase 1b/2 Trial Evaluating the Safety, Pharmacokinetics, and Efficacy of EP-104GI in Adults With Eosinophilic Esophagitis (RESOLVE)
Brief Title: A Trial to Evaluate EP-104GI in Adults With Eosinophilic Esophagitis (EoE).
Acronym: RESOLVE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eupraxia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP-104IAR-102 (RESOLVE)
Record Dates: First submitted 2022-10-19; First posted 2022-11-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- EP-104GI 4 mg (Experimental): 4 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 8 mg (Experimental): 8 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 20 mg (Experimental): 8 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 30 mg (Experimental): 12 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 48 mg (Experimental): 12 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 64 mg (Experimental): 16 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 80 mg (Experimental): 20 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 96 mg (Experimental): 16 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI 120 mg (Experimental): 20 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI Dose A or matching vehicle control (Placebo Comparator): 20 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI; Other: Matching vehicle control
- EP-104GI 160 mg (Experimental): 20 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI
- EP-104GI Dose B or matching vehicle control (Placebo Comparator): 20 submucosal injections of EP-104GI administered during an EGD procedure at the Baseline/Dosing visit.
  Interventions: Drug: EP-104GI; Other: Matching vehicle control

INTERVENTIONS:
Drug: EP-104GI — Extended-release fluticasone propionate [FP] for injectable suspension for gastrointestinal administration, Powder suspended in vehicle
Other: Matching vehicle control — A sterile liquid containing sterile water and excipients necessary to prepare a uniform suspension of the powder.
  Arms: EP-104GI Dose A or matching vehicle control; EP-104GI Dose B or matching vehicle control

SUMMARY:
A Phase 1b/2 study to explore the safety, efficacy and pharmacokinetics of EP-104GI in adults with eosinophilic esophagitis (EoE). Endoscopic and histologic assessments will also be evaluated to understand the local effects of EP-104GI on eosinophilic EoE disease activity. Approximately 27 to 33 participants will be enrolled in dose escalation: 3-6 participants per dose cohort. The number of participants enrolled in escalation will depend on the number of dose escalation cohorts evaluated, and dose cohorts needing to be expanded. An additional 10-24 participants will be enrolled in 1 or 2 cohorts of 10-12 participants each at tolerable dose regimen(s) selected based on the accumulated clinical data to identify the recommended phase 2 dose(s) (RP2D). In the Phase 2 randomized dose optimization portion of the study, approximately 120 subjects will be randomized to Dose A (120 mg total dose), Dose B (160 mg total dose), or matching vehicle control, with an overall assignment ratio of 1:1:1. The total number of participants in both portions of the study will be approximately 160. The study involves 8-10 site visits spread over approximately 52 weeks. Participants in an extended PK sub study will have up to 4 additional visits, to a maximum of 108 weeks post-dose. The participants will either receive the active study drug (EP-104GI) or matching vehicle control. Matching vehicle control will be used only in randomized dose optimization portion of the study. Participants randomized to receive vehicle control may receive EP-104GI (Dose A or Dose B) following the completion of Week 24 providing they meet eligibility criteria for crossover to EP-104GI. Participants randomized to receive EP-104GI on Day 0 will not receive EP-104GI or vehicle control at Week 24. The study drug or matching vehicle control will be administered by qualified personnel during an esophagogastroduodenoscopy (EGD) procedure at the Baseline/Dosing visit. Safety will be assessed throughout the study. Blood and urine samples will be collected at site visits for laboratory assessments and to measure plasma levels of EP-104GI. Participants will complete questionnaires to assess symptoms of dysphagia and odynophagia and will undergo 3-5 EGDs with esophageal biopsies at the Baseline, Week 4 (dose escalation phase only), Week 12, Week 24 (randomized dose optimization phase only), Week 26, and Week 52 (randomized dose optimization phase only).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic EoE;
* For women of childbearing potential, a negative pregnancy test and willing to use a highly effective method of birth control until end of study;
* Willing and able to adhere to study-related procedures and visit schedule;
* Willing and able to provide informed consent.

Criteria for crossover to EP 104GI from vehicle control (randomized dose optimization portion):

1. Has completed the randomized dose optimization portion of the trial to Week 24, inclusive
2. Without safety concerns for receiving EP 104GI ie, does not meet exclusion criteria or have other safety issue

Exclusion Criteria:

* Concomitant esophageal disease, relevant GI disease, or any condition, history, or laboratory abnormality that might interfere with the study;
* Oral or esophageal mucosal infection of any type (bacterial, viral, or fungal);
* Oropharyngeal or dental conditions that prevents normal eating;
* Severe esophageal motility disorders other than EoE;
* Contraindication to or factors that substantially increase risks associated with EGD or biopsy, or narrowing of the esophagus that precludes EGD with a standard 9-10 mm endoscope, stricture requiring dilation within 8 weeks prior to Screening, or the need for dilation prior to EGD at Baseline;
* Any condition for which the use of corticosteroids is contraindicated (Participants with well controlled non-insulin dependent diabetes are permitted);
* Active or quiescent systemic fungal, bacterial, viral, or parasitic infections, or ocular herpes simplex. Or recent use of IV or oral antibiotics;
* Hypersensitivity, or intolerance to corticosteroids, or to any of the ingredients in the investigational medicinal product, including carboxymethyl cellulose, and polysorbate 80, or to the ingredients in Synacthen / cosyntropin (used in the ACTH stimulation test);
* Recent use of disallowed medications, or unwillingness to not use disallowed medications during the study;
* Recent initiation of a elimination or elemental diet (dietary therapy must remain stable throughout the study);
* Morning serum cortisol level ≤ 5 μg/dL (138 nmol/L);
* Clinically significant abnormal laboratory values;
* Recent or currently planned participation in another interventional trial ;
* Previous participation in this study and had received study treatment;
* Females who are pregnant, breastfeeding, or planning to become pregnant during the study;
* Malignancies or history of malignancy within prior 5 years, except for treated or excised non-metastatic BCC, SCC of the skin, or cervical carcinoma in situ;
* History of alcohol or drug abuse;
* Any other reason, that, in the Investigator's opinion, unfavorably alters participant risk, confounds results, or prevents the participant from complying with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation- Incidence of treatment emergent adverse events (TEAEs) | 52 weeks
  TEAEs will be summarized by dose/cohort
Dose Escalation- Severity of treatment emergent adverse events (TEAEs) | 52 weeks
  TEAEs will be summarized by dose/cohort and severity (mild, moderate, severe).
Dose Escalation- Change from baseline in morning serum cortisol levels | 52 weeks
  Cortisol will be will be summarized by dose/cohort and over time and compared to pre-dose values. A prolonged and clinically significant reduction in cortisol may indicate adrenal insufficiency.
Dose Escalation- Plasma concentrations of fluticasone propionate | 108 weeks
  Plasma concentrations of fluticasone propionate over time will be used to calculate PK parameters for each dose/cohort.
Dose Escalation- Change from baseline in physical examination results, BMI and weight change. | 12 weeks
  Physical examination results, BMI and weight will be summarized by dose/cohort and over time and compared to pre-dose values.
Randomised Dose Optimization- Change from baseline in EoEHSS grade and stage scored in 3 regions of the esophagus within the injection area (proximal, mid, distal) | 24 weeks
  The EoEHSS scores the stage and grade of 8 histologic items: eosinophil inflammation, basal zone hyperplasia, dilated intercellular spaces, eosinophil abscesses, surface layering, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis), on separate 4-point Likert scales. A composite EoEHSS grade and stage scores are calculated by summing the individual grade and stage items and dividing by the maximum score for evaluated items (range, 0-1). A lower score indicates improvement.

SECONDARY OUTCOMES:
Dose Escalation- Peak eosinophil count (PEC) | 36 weeks
  Biopsy specimens will be used to evaluate peak eosinophil counts (PEC). A higher number of eosinophils indicates more severe histological disease.
Dose Escalation- Change from baseline in the Straumann Dysphagia Index (SDI) score | 52 weeks
  The SDI is a patient-reported outcome measure of dysphagia with a 7-day recall period. The SDI assesses the frequency and intensity of dysphagia on two separate 5-point and 6-point scales. Total SDI scores are calculated by adding the two sub-scores (range, 0-9), with a higher total score indicating more severe dysphagia.
Dose Escalation- Change from baseline in dysphagia measured on an 11 point Likert scale | 52 weeks
  The participant will assess the severity of their dysphagia symptoms (troubles to swallow) over the previous 7-days using an 11-point Likert scale where 0 = no trouble and 10 = most severe trouble swallowing.
Dose Escalation- Change from baseline in the EoE Endoscopic Reference Score (EREFS) | 36 weeks
  Endoscopic Reference Score (EREFS) scoring system is used to determine the severity of 5 endoscopic findings: edema, rings, exudates, furrows, and strictures. The total EREFS is calculated by summing the grades of the 5 individual endoscopic items (range, 0 to 9), with higher scores indicating more severe endoscopic disease.
Dose Escalation- Change from baseline in odynophagia measured on an 11 point Likert scale | 52 weeks
  The participant will assess the severity of their pain during swallowing over the previous 7 days using an 11 point Likert scale where 0 = no pain and 10 = most severe pain during swallowing.
Dose Escalation- Change from baseline in EoE Histology Scoring System (EoEHSS) score | 36 weeks
  The EoEHSS scores the stage and grade of 8 histologic items: eosinophil inflammation, basal zone hyperplasia, dilated intercellular spaces, eosinophil abscesses, surface layering, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis), on separate 4-point Likert scales. A composite EoEHSS grade and stage scores are calculated by summing the individual grade and stage items and dividing by the maximum score for evaluated items (range, 0-1). A lower score indicates improvement.
Randomised Dose Optimization- Change from baseline in the Straumann Dysphagia Index (SDI) score | 52 weeks
  The SDI is a patient-reported outcome measure of dysphagia with a 7-day recall period. The SDI assesses the frequency and intensity of dysphagia on two separate 5-point and 6-point scales. Total SDI scores are calculated by adding the two sub-scores (range, 0-9), with a higher total score indicating more severe dysphagia.
Randomised Dose Optimization- Change from baseline in the Dysphagia symptom questionnaire (DSQ) v4.0 and "Dysphagia days" | 52 weeks
  The DSQ is assessed daily over a period of 14 days and comprises four questions; one question on whether the participant has eaten solid food and three questions on the presence and severity of EoE dysphagia."Dysphagia Days" is defined as the number of days with a yes answer to the following question: During any meal today, did food go down slowly or get stuck in your throat or chest?
Randomised Dose Optimization- Change from baseline in the Eosinophilic Esophagitis Impact Questionnaire (EoE IQ) | 52 weeks
  The EoE-IQ is a validated PRO instrument consisting of 11 questions assessing the impact of EoE on health related quality of life.
Randomised Dose Optimization- Change from baseline in the Patient Global Impression of Change (PGIC) | 52 weeks
  The PGIC reflects a participant's belief about the efficacy of treatment on a 7 point scale rating on a 4 point scale.
Randomised Dose Optimization- Change from baseline in the Patient Global Impression of Severity (PGIS) | 52 weeks
  The PGIS reflects a participant's belief about the efficacy of treatment based on severity ranging from none to very severe.
Randomised Dose Optimization- Change from baseline in peak eosinophil count (PEC) | 52 weeks
  Biopsy specimens will be used to evaluate peak eosinophil counts (PEC). A higher number of eosinophils indicates more severe histological disease.
Randomised Dose Optimization- Change from baseline in the EoE Endoscopic Reference Score (EREFS) in 3 regions of the esophagus within the injection area (proximal, mid, distal) | 52 weeks
  Endoscopic Reference Score (EREFS) scoring system is used to determine the severity of 5 endoscopic findings: edema, rings, exudates, furrows, and strictures. The total EREFS is calculated by summing the grades of the 5 individual endoscopic items (range, 0 to 9), with higher scores indicating more severe endoscopic disease.
Randomised Dose Optimization- Change in endoscopist's global impression of severity | 52 weeks
  The PGIC reflects a participant's belief about the efficacy of treatment on a 7 point scale rating overall improvement; the PGIS reflects a participant's belief about the severity of their symptoms on a 4 point scale
Randomised Dose Optimization- Change from baseline in EoE Histology Scoring System (EoEHSS) score in 3 regions of the esophagus within the injection area (proximal, mid, distal), excluding Week 24 as this is the primary endpoint | 52 weeks
  The EoEHSS scores the stage and grade of 8 histologic items: eosinophil inflammation, basal zone hyperplasia, dilated intercellular spaces, eosinophil abscesses, surface layering, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis), on separate 4-point Likert scales. A composite EoEHSS grade and stage scores are calculated by summing the individual grade and stage items and dividing by the maximum score for evaluated items (range, 0-1). A lower score indicates improvement.
Randomised Dose Optimization- Change from baseline in morning serum cortisol levels | 52 weeks
  Cortisol will be will be summarized by dose/cohort and over time and compared to pre-dose values. A prolonged and clinically significant reduction in cortisol may indicate adrenal insufficiency.
Randomised Dose Optimization- Change from baseline in vital signs (temperature, blood pressure, pulse, and respiratory rate) results | 52 weeks
  Vital signs (temperature, blood pressure, pulse, and respiratory rate) results will be summarized by dose/cohort and over time and compared to pre-dose values.
Randomised Dose Optimization- Change from baseline in physical examination results, BMI and weight change. | 52 weeks
  Physical examination results, BMI and weight will be summarized by dose/cohort and over time and compared to pre-dose values.
Randomised Dose Optimization- Plasma concentrations of fluticasone propionate | 108 weeks
  Plasma concentrations of fluticasone propionate over time will be used to calculate PK parameters for each dose/cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kowalski, MD PhD, Study Director — Eupraxia Pharmaceuticals
Locations (19):
- Australia (9):
  - Campbelltown Private Hospital, Sydney, New South Wales
  - Mater Hospital Brisbane, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Coastal Digestive Health, Maroochydore, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Health Box Hill, Box Hill, Victoria
  - Northern Hospital Epping, Epping, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - UoA - South Edmonton Gastroenterology Research Clinic, Edmonton, Alberta
  - G.I. Research Institute, Vancouver, British Columbia
  - McGill University Health Center, Montreal, Quebec
- Amsterdam UMC, Amsterdam, Netherlands
- New Zealand (2):
  - Aotearoa Clinical Trials, Papatoetoe, Auckland
  - Capital Coast and Hutt, Lower Hutt
- Universitätsspital Zürich, Zurich, Switzerland
- United Kingdom (2):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Cardiff and Vale University Health Board-Wales, Cardiff

IPD SHARING:
Plan to Share IPD: No